CLINICAL TRIAL: NCT06274424
Title: Association Between Hair Cortisol and Symptoms in Children With Psychopathology During CBT
Brief Title: Hair Cortisol and Symptoms in Children With Psychopathology During CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Sarianna Barron-Linnankoski, Principal Investigator, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/211/2016 and HUS/2699/2018
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Child Behavior Problem
Keywords: Children; group cognitive behavioral therapy; hair cortisol concentration; internalizing symptoms; externalizing symptoms; sleep disturbance symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Cognitive Behavioral Therapy Intervention (Experimental): The Friends Program
  Interventions: Behavioral: The Friends Program

INTERVENTIONS:
Behavioral: The Friends Program — A group CBT intervention comprising ten weekly 60-minute sessions followed by two booster sessions.

SUMMARY:
This study aims to examine the relationship between hair cortisol concentration and behavior and sleep disturbance symptoms in children with psychiatric disorders. It also investigates potential changes in hair cortisol and symptomatology after group-based cognitive behavior therapy. Furthermore, the study explores the effects of any alterations in hair cortisol concentration levels on potential behavior and sleep disturbance symptom change over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of anxiety or depression
* deficiencies in emotional and behavioral skills impairing functioning
* sufficient social and cognitive skills to participate in group work.

Exclusion Criteria:

* excessive physical aggression
* excessive physical restlessness
* severity of psychiatric symptoms requiring individual psychotherapy (e.g., acute suicidality).

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Hair Cortisol Concentration | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Level of hair cortisol concentration measured from hair samples
Parent- and teacher rated internalizing and externalizing symptoms | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  The Achenbach System of Empirically Based Assessment (ASEBA). Scores below 60 reflect the normal range, scores from 60 to 63 the borderline range, and scores above 63 the clinical range
Child-rated internalizing symptoms | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  The Spence Children´s Anxiety Scale. A total score of 60 or higher is indicative of elevated anxiety.
Parent-rated sleep disturbance symptoms | Before and after the group cognitive behavioral intervention (duration from pre-GCBT to post-GCBT circa 4.7 months), and at a 7-month follow-up
  Sleep Disturbance Scale for Children (SDSC). A cutoff score of 39 and above has been suggested to identify children with sleep disturbance.

IPD SHARING:
Plan to Share IPD: No